CLINICAL TRIAL: NCT01738789
Title: European Multicenter Validation of an ADNEXMR SCORING System for Characterizing Adnexal Masses: "EURAD-MR Classification"
Brief Title: EURAD-MR Classification : European Multicenter Study
Acronym: EURAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Société d'Imagerie de la Femme (Other)
Responsible Party: Principal Investigator, Isabelle Thomassin-Naggara, Full Professor, Société d'Imagerie de la Femme
Other Study IDs: SIFEM-2013-1
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Tumor
Keywords: Adnexal masses; Magnetic resonance imaging; Ovarian tumor
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An adnexal mass is the most common indication for gynaecological surgery . Pre operative characterization is crucial and a scoring system would be useful to standardize the imaging report and thus, improve patient management. Recently, our center developed the first MR scoring system named ADNEXMR SCORING system in a retrospective study which is accurate and reproducible (1). Our objectives are to perform an external prospective validation of this scoring system, to evaluate its potential impact on therapeutic strategy and to test its reproducibility.

This is a prospective large multicenter study. All patients with a sonographically indeterminate adnexal mass referred for MR imaging will be consecutively included in each center. Then, patients will undergo a routine pelvic MR imaging. Prospectively, one senior and one junior radiologists independently analyze the different MR criteria to characterize adnexal masses. The MR report will be issued as standard and the patient will be managed accordingly. Then, the reader will classify the mass using ADNEXMR SCORING system. The classification will be compared to the reference standard as defined below. The reproducibility of the classification will be tested between the junior and the senior radiologist. After anonymisation, images will be analyzed by another senior radiologist of another center blinded from any clinical or ultrasonographical data and correlated with the reference standard.

Reference standard: Reference standard will be surgical procedure with histology or standard clinical follow-up depending on most appropriate routine practice.

Sample size: The sample size was computed to ensure a power of at least 90% (with a two-sided type I error rate of 5%) to conclude that SCORE 2 and 3 and SCORE 4 and 5 would have a different PPV. It would thus be necessary to have at least 569 patients classified as SCORE 2, 259 as SCORE 3, 52 as SCORE 4 and 51 as SCORE 5 (18). Given the prevalences, and assuming 6% of patients would be classified, as SCORE 1 and 10% would be lost to follow-up, 1340 patients will be included in this study to insure a probability of at least 95% to obtain the aforementioned number of patients in each score category. The inclusion period will last 18 months (extension for a period of 12 months) and monitoring will continue for 2 years.

Thomassin Naggara I., et al. Development and preliminary validation of an MRI Scoring system for Adnexal Masses. Radiology 2013, May;267(2):432-43.

DETAILED DESCRIPTION:
All patients with an indeterminate ultrasonographically adnexal mass referred for MR imaging will be consecutively included in each center.

Inclusion Criteria

* Patient ≥ 18 years old
* With indeterminate ultrasonographic adnexal mass
* Informed consent

Non inclusion Criteria

* Pregnant women
* Pacemaker, ferromagnetic materials, or foreign body at risk of mobilization
* Intolerance to iodinated or gadolinium contrast agents, or severe renal insufficiency (GFR <30 ml/min/1.73m²).

Objectives • Primary objective: Evaluate if ADNEXMR SCORING system is relevant for reporting pelvic magnetic resonance imaging (MRI) examinations performed for characterization of sonographically indeterminate adnexal masses in an external prospective multicenter study

• Secondary objectives and endpoints: Evaluate

1. The potential impact of applying the score to the therapeutic strategy, in particular to measure the possible reduction in oncologic surgery in benign cases
2. If ADNEXMR SCORING system improves reproducibility of MR report for characterization of adnexal masses
3. If ADNEXMR SCORING system is as accurate if the radiologist is blinded from any clinical and ultrasonographic data

Main endpoint Joint analysis of true negative and false negative rates according to ADNEXMR SCORING system as compared to the histological results (or follow-up outcome, see "reference standard", below) with an evaluation of the sensitivity and the specificity of the score

ELIGIBILITY:
Inclusion Criteria

* Patient ≥ 18 years old
* With sonographically indeterminate adnexal mass
* Informed consent

Exclusion Criteria

* Pregnant women (relative contra indication for gadolinium injection)
* Pacemaker, ferromagnetic materials, or foreign body at risk of mobilization or any other contra-indication to MR imaging.
* Intolerance to iodinated or gadolinium contrast agents, or severe renal insufficiency (GFR <30 ml/min/1.73m²).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a sonographically indeterminate adnexal mass referred for MR imaging will be consecutively included in each center
Sampling Method: Probability Sample
Enrollment: 1340 (Actual)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
External validation of Adnex MR scoring system | 24 months
  Evaluate if ADNEXMR SCORING system is relevant for reporting pelvic magnetic resonance imaging (MRI) examinations performed for characterization of sonographically indeterminate adnexal masses in an external prospective multicenter study

SECONDARY OUTCOMES:
Potential reduction of unnecessary surgery | 24 months
  The potential impact of applying the score to the therapeutic strategy, in particular to measure the possible reduction in unnecessary surgery in benign cases
Reproducibility of the score | 24 months
  If ADNEXMR SCORING system improves reproducibility of MR report for characterization of adnexal masses
Comparison between a blinded and an unblinded radiologist regarding sonographic data | 24 months
  If ADNEXMR SCORING system is as accurate if the radiologist is blinded from any clinical and ultrasonographic data

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Thomassin-Naggara, MD, PhD, Study Chair — Assistance Publique des Hopitaux de Paris, Université Pierre et Marie Curie; Andrea Rockall, MD, Study Director — Imperial College of London; Marc Bazot, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (24):
- University Institute of Radiology, Salzburg, Austria
- University Hospital Dubrav, Zagreb, Croatia
- France (12):
  - Centre Oscar Lambret, Lille
  - Hopital de la Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hopital de Lapeyronie, Montpellier
  - Tenon Hospital, Paris
  - Centre imagerie Pyramides, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Hopital Lariboisière, Paris
  - Hôpital de la Pitié-Salpétrière, Paris
  - Institut Curie - Huguenin, Paris
  - Hopital de Valenciennes, Valenciennes
  - Institut Gustave Roussy, Villejuif
- Umberto I hospital Sapienza, Roma, Italy
- Portugal (2):
  - Hospital da Luz, Lisbon
  - Instituto Portuges de Oncologia de Lisboa Francisco Gentil, Lisbon
- Clinical Center of Vojvodine, Novi Sad, Serbia
- University Hodpital Dubrav, Baden, Switzerland
- United Kingdom (5):
  - Addenbrokes hospital, Cambridge
  - Barts Health NHS trust, London
  - Imperial College Healthcare, London
  - University College London, London
  - Steeping Hill hospital, Stockport

REFERENCES:
- [Derived] Wengert GJ, Dabi Y, Kermarrec E, Jalaguier-Coudray A, Poncelet E, Porcher R, Thomassin-Naggara I, Rockall AG; EURAD Study Group. O-RADS MRI Classification of Indeterminate Adnexal Lesions: Time-Intensity Curve Analysis Is Better Than Visual Assessment. Radiology. 2022 Jun;303(3):566-575. doi: 10.1148/radiol.210342. Epub 2022 Mar 1. PMID 35230183